CLINICAL TRIAL: NCT06862219
Title: A Multicenter, Phase 4, Open-label, Single-arm, Safety Study of Enfortumab Vedotin in Adult Indian Participants With Previously Treated Locally Advanced or Metastatic Urothelial Cancer
Brief Title: A Safety Study of Enfortumab Vedotin in Indian Adults With Urothelial Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7465-CL-4001
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Urothelial Carcinoma
Keywords: PADCEV; ASG-22CE; Urothelial cancer; Enfortumab Vedotin
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Enfortumab Vedotin (EV) - All participants (Experimental): Participants will receive enfortumab vedotin (EV) on days 1, 8 and 15 of each 28 day cycle
  Interventions: Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Enfortumab Vedotin — Intravenous Infusion
  Other Names: ASG-22CE; PADCEV

SUMMARY:
This study is for Indian adults in India who have cancer in the bladder lining (urothelial cancer). Their cancer is advanced or has spread to other parts of the body. Enfortumab vedotin is a treatment for this type of cancer.

The main aim of the study is to confirm the safety of enfortumab vedotin in Indian adults with urothelial cancer.

During the study, people will receive enfortumab vedotin. The study treatment will be given to people slowly through a tube into a vein. This is called an infusion. People will receive 3 separate infusions of enfortumab vedotin in each 28-day (4 weeks) treatment cycle.

People visit their study clinic for health-checks several times during and after they receive enfortumab vedotin.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically confirmed urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter or urethra). Participants with urothelial carcinoma (transitional cell) with squamous differentiation or mixed cell types are eligible.
* Participant must have experienced radiographic progression or relapse during or after a checkpoint inhibitor (CPI) (anti-PD-1 or anti-PD-L1) for locally advanced (LA) or metastatic disease. Participants who discontinued CPI treatment due to toxicity are eligible provided that they have evidence of disease progression following discontinuation. The CPI need not be the most recent therapy. Participants for whom the most recent therapy has been a non-CPI based regimen are eligible if they have progressed / relapsed during or after their most recent therapy. LA disease must not be amenable to resection with curative intent.
* Participant must have received a platinum-containing regimen (cisplatin or carboplatin) in the metastatic / LA, neoadjuvant or adjuvant setting. If platinum was administered in the ajuvant/neoadjuvant setting, the participant must have progressed within 12 months of completion.
* Participant must have measurable metastatic or LA disease at baseline according to RECIST version 1.1.
* Participant has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant's baseline laboratory data meets protocol specified of criteria.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who has a negative urine or serum pregnancy test at screening or within 7 days prior to day 1 and agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after final study intervention administration.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for approximately 6 months after final study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 6 months after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 6 months after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 6 months after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 6 months after final study intervention administration.
* Participant agrees not to participate in another interventional study while receiving study intervention in the present study.

Exclusion Criteria:

* Participant has preexisting sensory or motor neuropathy grade ≥ 2.
* Participant has active central nervous system (CNS) metastases. Participant with treated CNS metastases is permitted on study if all the following are true:

  * CNS metastases have been clinically stable for at least 6 weeks prior to screening
  * If requiring steroid treatment for CNS metastases, the participant is on a stable dose ≤ 20 mg/day of prednisone or equivalent for at least 2 weeks
  * Baseline scans show no evidence of new or enlarged brain metastasis
  * Participant does not have leptomeningeal disease
* Participant has ongoing clinically significant toxicity (grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery).

  * Participant with ≤ grade 2 immunotherapy-related hypothyroidism or panhypopituitarism may be enrolled when well-maintained / controlled on a stable dose of hormone replacement therapy (HRT) (if indicated).
  * Participant with ongoing ≥ grade 3 immunotherapy-related hypothyroidism or panhypopituitarism are excluded.
  * Participant with ongoing immunotherapy-related colitis, uveitis, myocarditis or pneumonitis, or participant with other immunotherapy-related AEs requiring high doses of steroids (> 20 mg/day of prednisone or equivalent) are excluded.
* Participant has history of another malignancy within 3 years before the first dose of study intervention or any evidence of residual disease from a previously diagnosed malignancy.

  * Participant with non-melanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low-risk (per standard guidelines) localized prostate cancer under active surveillance / watchful waiting without intent to treat, or carcinoma in situ of any type (if complete resection was performed) are allowed.
* Participant with a positive hepatitis B surface antigen and/or anti-hepatitis B core antibody and a negative polymerase chain reaction assay at baseline should receive appropriate antiviral prophylaxis or regular surveillance monitoring as per local or institutional guidelines.
* Participant has active hepatitis C infection or known human immunodeficiency virus infection. Participant who has been treated for hepatitis C infection is permitted if they have documented sustained virologic response of ≥ 12 weeks.
* Participant has documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III to IV within 6 months prior to the first dose of study intervention administration.
* Participant has known active keratitis or corneal ulcerations. Participant with superficial punctate keratitis is allowed if the disorder is being adequately treated.
* Participant has other underlying medical condition that would impair the ability of the participant to receive or tolerate the planned treatment and follow-up.
* Participant has history of uncontrolled diabetes mellitus within 3 months of the first dose of study intervention. Uncontrolled diabetes is defined as HbA1c ≥ 8 percent or HbA1c between 7 percent and < 8 percent with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Participant has prior treatment with enfortumab vedotin or other monomethyl auristatin E (MMAE)-based antibody drug conjugate (ADCs).
* Participant is currently receiving systemic antimicrobial treatment for viral, bacterial, or fungal infection at the time of first dose of enfortumab vedotin. Routine antimicrobial prophylaxis is permitted.
* Participant has radiotherapy or major surgery within 4 weeks prior to first dose study intervention administration.
* Participant has had chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy that is not completed 2 weeks prior to first dose of study intervention administration.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to enfortumab vedotin or to any excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate, and polysorbate 20); OR participant has known hypersensitivity to biopharmaceuticals produced in CHO cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events | Up to 8 months
  Adverse events (AE) will be coded using MedDRA. An AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Number of participants with laboratory value abnormalities and/or AEs | Up to 7 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to 7 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 6.5 months
  Number of participants with potentially clinically significant ECG values.
Number of Participants at each grade of Eastern Cooperative Oncology Group (ECOG) Performance Status score | Up to 7 months
  The ECOG scale will be used to assess performance status. Scores range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Confirmed Overall Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST V1.1) per investigator assessment | Up to 34 months
  ORR is defined as the proportion of participants whose best overall response is a confirmed complete response (CR) or partial response (PR) according to RECIST version 1.1 per investigator assessment
Duration of Response (DOR) according to RECIST version 1.1 per investigator assessment | Up to 34 months
  DOR is defined as the time from the date of the first documented response (CR or PR that is subsequently confirmed) per RECIST version 1.1 as determined by investigator to the date of first documented radiological disease progression per RECIST version 1.1 or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (8):
- India (8):
  - Site IN91016, New Delhi, National Capital Territory of Delhi
  - Site IN91017, Dumas, Surat
  - Site IN91005, Varanasi, Uttar Pradesh
  - Site IN91012, Ahmedabad
  - Site IN91010, Bhubaneswar
  - Site IN91008, Mumbai
  - Site IN91009, Nagpur
  - Site IN91001, Surat

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/